CLINICAL TRIAL: NCT05931744
Title: The Role of Budesonide Intrapolyp Injection in the Management of Type 2 Chronic Rhinosinusitis . A Randomized Clinical Trial
Brief Title: The Role of Budesonide Intrapolyp Injection in the Management of Type 2 Chronic Rhinosinusitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ibrahim M. Gehad, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKSU 50-7-8
Record Dates: First submitted 2023-05-12; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: CRSwNP; Intranasal steroid injection; Budesonide
MeSH Terms: interventions — Budesonide; Prednisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral steroid (Active Comparator): patients given prednisone 1 mg/kg for 3 days then tapered by 5mg daily for two weeks
  Interventions: Drug: Prednisone
- Budesonide Intrapolyp injection (Experimental): patients given budesonide 0.5 mg/2ml intrapolyp injection once weekly for 5 consecutive weeks
  Interventions: Drug: Budesonide
- Saline intrapolyp injection (Placebo Comparator): patients given 2ml normal saline intrapolyp injection once weekly for 5 consecutive weeks
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Budesonide — after application of topical vasoconstrictor packs into both nasal cavities, using 1 cc 28 gauge needle sterile syringe, one pack of budesonide ampule 0.5 mg/2ml was injected into visible polyps on both cavities 1 ml in each cavity weekly for 5 consecutive weeks
  Arms: Budesonide Intrapolyp injection
Drug: Prednisone — patients given oral prednisone 1 mg/ kg with max. dose 70 mg/d divided into two doses for 3 days then tapered gradually for two weeks
  Arms: Oral steroid
Drug: Saline — saline intrapolyp injection
  Arms: Saline intrapolyp injection

SUMMARY:
To investigate the usage of budesonide as an agent in the injection of Type 2 chronic rhinosinusitis with nasal polyps

DETAILED DESCRIPTION:
this is a randomized controlled clinical trial where 3 groups with nasal polyps will be treated medically, Group A with oral corticosteroids, Group B with budesonide intrapolyp injection, Group C with placebo saline intrapolyp injection

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 2 CRSwNP -
* elevated serum IgE & high absolute eosinophilia
* with any grade of nasal polyps
* ages between 18 and 60 years old
* patients who didn't have any contraindications of systemic steroids

Exclusion Criteria:

* All patients with previous nasal surgeries
* All patients with cystic fibrosis, ciliary dyskinesia, antrochoanal polyp, fungal sinusitis, unilateral nasal polyps, nasal tumors,
* patients who took systemic steroids in the last 6 months before our study
* patients with any previous nasal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Sino-Nasal Outcome Test "SNOT-22" Score | 6 months
  subjective method to assess the patient's quality of life "QOL" and the severity of the disease before and after treatment, The lower the score, The better the condition
CT Lund Mackay | 6 months
  the radiological evaluation of patients with nasal polyps where each sinus was solitarily assigned a score from (0 to 2), where the Osteomeatal Complex was given only (0 or 2), each side was evaluated on its own and the sum of all sinuses was calculated. A combined score of 24 was the maximum. Investigators asked the patients for a CT scan before starting the treatment and 3 months after the completion of each treatment protocol
Total nasal Polyp score "TNPS" | 6 months
  the clinical assessment of nasal polyps, the total nasal polyp score "TNPS" was used where polyp size was evaluated through endoscopy and given a score from (0 to 3). TNPS was calculated as the sum of the score on each side, and patients were assessed on regular visits before receiving treatment, 1 week after treatment, and after 3 months
Serum IgE | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University hospital, Kafrelsheikh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes